CLINICAL TRIAL: NCT03694652
Title: Text Messaging to Promote Mobility in Overweight/Obese Adults With Peripheral Artery Disease
Brief Title: Texting for Mobility in Overweight/Obese Adults With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00141458; 1R56HL138244 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-02

CONDITIONS: Overweight and Obesity
Keywords: Text messaging; PAD
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet; Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE+DApp (Experimental): Participants in this group will receive combined intervention and a mobile phone app.
  Interventions: Behavioral: PACE; Behavioral: Diet; Other: App
- PACE+Dface-to-face (Active Comparator): Participants in this group will receive combined intervention and in person/phone communication.
  Interventions: Behavioral: PACE; Behavioral: Diet; Other: Face-to-face

INTERVENTIONS:
Behavioral: PACE — Patient-centered Assessment and Counseling for Exercise [PACE] program
Behavioral: Diet — Motivating healthy dietary habits
Other: App — Using an app to deliver communication to the participant.
  Arms: PACE+DApp
Other: Face-to-face — Using in person meetings and/or phone communication with the participant.
  Arms: PACE+Dface-to-face

SUMMARY:
By doing this study, researchers hope to learn about the feasibility of using a mobile application to help overweight or obese adults with PAD increase their walking distance and lose weight.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) or poor leg circulation affects 8 to 12 million Americans including non-Hispanic Whites, African Americans and Latinos. Having PAD can limit how far you can walk. Many patients with PAD are also overweight or obese. Weight loss among overweight or obese adults with PAD may improve walking distance. Given how common obesity or being overweight is among persons with PAD, interventions are needed to address weight loss in this population.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (body mass index >=27 kg/m2)
* Have symptomatic PAD
* English speaking
* Have 24 hour access to a cell phone

Exclusion Criteria:

* Cannot tolerate fruits and vegetables, fiber, and/or a low fat diet, as informed by a physician and/or registered dietician
* Restricted intake of water
* Pregnancy
* Prior major amputation (foot or lower leg) or critical leg ischemia (tissue loss, gangrene, or ulcers)
* Use of supplemental oxygen
* Heart attack within preceding 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracie C Collins, MD, MPH, MHCDS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas School of Medicine, Wichita, Kansas, United States

REFERENCES:
- [Derived] Collins T, Geana M, Overton K, Benton M, Lu L, Khan F, Rohleder M, Ahluwalia J, Resnicow K, Zhu Y. Use of a Smartphone App Versus Motivational Interviewing to Increase Walking Distance and Weight Loss in Overweight/Obese Adults With Peripheral Artery Disease: Pilot Randomized Trial. JMIR Form Res. 2022 Feb 3;6(2):e30295. doi: 10.2196/30295. PMID 35113020

RESULTS

PARTICIPANT FLOW:
Groups:
- PACE+DApp: Participants in this group will receive a physical activity and dietary intervention via a mobile phone app.
  PACE: Patient-centered Assessment and Counseling for Exercise [PACE] program to promote physical activity
  Diet: Motivating healthy dietary habits
  App: Using an app to deliver communication to the participant.
- Motivational Interviewing: Participants in this group will receive motivational interviewing - in-person and via telephone.
  Motivational Interviewing: Motivational interviewing counseling is used to promote physical activity and healthy dietary habits.
Period: Overall Study
Arm/Group | PACE+DApp | Motivational Interviewing
Started | 13 | 16
Completed | 11 | 14
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- PACE+DApp: Participants in this group will receive a physical activity and dietary intervention via a mobile phone app.
  PACE: Patient-centered Assessment and Counseling for Exercise [PACE] program to motivate physical activity
  Diet: Motivating healthy dietary habits
  App: Used to deliver the interventions
- Motivational Interviewing: Participants in this group will receive counseling - motivational interviewing.
  Motivational interviewing was used to motivate physical activity and health dietary habits
  MI was delivered face-to-face initially followed by telephone for subsequent sessions (total sessions were 5)
- Total: Total of all reporting groups
Arm/Group | PACE+DApp | Motivational Interviewing | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.12 (8.34) | 68.39 (7.36) | 66.03 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 14 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Walking Distance
Description: Walking distance as measured by the 6 minute walk test.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: meters
Groups:
- PACE+DApp: Participants in this group will receive combined intervention via a mobile phone app.
  PACE: Patient-centered Assessment and Counseling for Exercise [PACE] program was used to motivate physical activity
  Diet: health dietary habits (reducing sodium, increasing fruits and vegetables, increasing whole grains, mindful eating, decreasing sugary drinks)
  App: The app was used to deliver both physical activity and healthy dietary habits.
- Motivational Interviewing: Participants in this group will receive counseling (motivational interviewing) an initial face-to-face session followed by four phone sessions.
  Motivational interviewing was used to promote physical activity and healthy dietary habits.
Arm/Group | PACE+DApp | Motivational Interviewing
Number analyzed (Participants) | 11 | 14
meters | 331.19 (58.63) | 298.67 (101.20)

2. Secondary Outcome: Weight Loss
Description: Change in weight, collected at two time points.
Time Frame: Month 3
Measure: Mean (95% Confidence Interval); unit: lbs.
Arm/Group | PACE+DApp | Motivational Interviewing
Number analyzed (Participants) | 11 | 14
lbs. | 2.3 [0.7 to 3.4] | 10.1 [3.0 to 17.9]

3. Secondary Outcome: Quality of Life (QoL)
Description: QoL as measured by the Vascular Quality of Life Questionnaire. There are 25 questions that are each scored 1-7. The total score is determined by all adding the score from each of the 25 questions and dividing by 25. The total range is 1-7 and a higher score indicates a better quality of life.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: units on a scale;
Arm/Group | PACE+DApp | Motivational Interviewing
Number analyzed (Participants) | 11 | 14
units on a scale; | 5.09 (1.37) | 5.36 (0.75)

4. Secondary Outcome: Physical Activity
Description: Physical activity to be measured using the Exercise Behavior Questionnaire from the Stanford Patient Education Research Center. Scores are for type of activity, length of activity, time spent in aerobic activities, and an assessment of time spent in stretching and strengthening exercises. For the manuscript, we only focused on aerobic activity and we did not include stretching or strengthening exercise scores.
  Participants were asked how often during the past week they performed aerobic exercises on a scale of 0 (none) to 4 (more than 3 hours per week). Scores were converted by the overall time spent in aerobic exercises per week and range from 0 to 180 with higher scores indicating more time spent doing aerobic exercises.
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PACE+DApp | Motivational Interviewing
Number analyzed (Participants) | 11 | 14
units on a scale | 22.73 (16.56) | 27.32 (27.18)

5. Secondary Outcome: Dietary Habits
Description: Dietary habits tracked using the Fat-Related Diet Habits Questionnaire. Questions were rated on a 4-point scale, where 1 indicates healthy and 4 less healthy eating habits. The questionnaire included ﬁve sections (i) replacing high fat foods with low fat substitutes (score range: 7-28); (ii) modifying high fat foods (range: 3-12); (iii) avoiding high fat cooking methods (score range: 4-16); (iv) consumption of fresh fruit and vegetables as a snack (score range: 3-12); and (v) choosing specially manufactured low fat food (score range: 5-20). The total score is calculated from the sum of section scores divided by 5 (range from 4.4 to 17 with higher scores representing more unhealthy eating habits)
Time Frame: Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PACE+DApp | Motivational Interviewing
Number analyzed (Participants) | 11 | 14
score on a scale | 2.61 (0.32) | 2.45 (0.52)

ADVERSE EVENTS:
Time Frame: three months
Arm/Group | PACE+DApp | Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03694652/Prot_SAP_000.pdf